CLINICAL TRIAL: NCT04355585
Title: Revisiting the Mechanism of the Anti-inflammatory Effect of Colchicine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Lindsey R. Baden, MD, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020P000440
Record Dates: First submitted 2020-04-18; First posted 2020-04-21 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Colchicine Mechanism of Action
Keywords: pharmacology
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Stratified randomization according to sex will be performed. Each group will be randomized to receive colchicine or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study in which investigators, participants, site personnel, and laboratory staff will be blinded during the study. Only the research pharmacy will have access to randomization and treatment assignments.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Male (Experimental): Participants in this group will be randomized to receive either a single dose of colchicine (1.8mg administered over 1 hour in the form of tablets) or placebo.
  Interventions: Drug: Colchicine Tablets; Drug: Placebo oral tablet
- Female (Experimental): Participants in this group will be randomized to receive either a single dose of colchicine (1.8mg administered over 1 hour in the form of tablets) or placebo.
  Interventions: Drug: Colchicine Tablets; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Colchicine Tablets — 1.8mg of Colchicine given over 1 hour (1.2 mg followed by 0.6 mg 1 hour later)
Drug: Placebo oral tablet — Placebo given over 1 hour (first tablet followed by second tablet 1 hour later)

SUMMARY:
We are doing this research study to better understand the mechanism of action of colchicine, a drug commonly prescribed for gout. Precisely, we aim to evaluate the effect of colchicine on a specific protein (GDF15) blood levels at different timepoints after its administration.

This research study will compare GDF15 blood levels after the administration of colchicine or placebo. The placebo looks exactly like colchicine but contains no active drug. During this study, participants may get a placebo instead of colchicine. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

DETAILED DESCRIPTION:
This will be a randomized, placebo-controlled, double-blind, pilot study evaluating the effect of a single FDA-approved dose of colchicine in healthy adults on plasma GDF15 levels. Randomization will be stratified by sex as this may be a factor influencing GDF15 levels.

On Day 1, subjects will be admitted on the CCI 9A unit early in the morning, 30 minutes before the study drug administration. They will be asked to fast from midnight before the dose until 2 hours after. Water is allowed during the fasting period. Baseline blood tests will be drawn and a peripheral line will be left in place for further blood draws. A dose of either colchicine or placebo will be administered. Blood samples will be drawn at 2, 4, 6, 8, 10 and 12 hours. The patient will be discharged home after the last blood draw and the removal of the peripheral line. Two other blood draws will be performed using standard procedures at 24 and 48 hours post study drug administration at the research clinic

ELIGIBILITY:
Inclusion Criteria:

* Participant able to understand and sign the informed consent of the study
* Healthy male or female aged from 18 to 50 years.
* Participant considered healthy after evaluation such as medical history and screening laboratories.

Exclusion Criteria:

* Pregnant or lactating women
* Use of colchicine within 28 days prior to study drug administration.
* Renal insufficiency (GFR < 50 mL/min)
* Use of any drug or product known to interact with colchicine including CYP3A4 and/or P-glycoprotein (P-gp) inhibitors in the 14 days prior study drug administration, such as atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, amprenavir, aprepitant, diltiazem, erythromycin, fluconazole, fosamprenavir, verapamil, cyclosporine and ranolazine. Significant consumption of grapefruit juice can also inhibit CYP3A4. Interactions may also be seen with fibrates (e.g., gemfibrozil), HMG-CoA reductase inhibitors (statins) and digoxin.
* History of colchicine allergy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Plasma GDF15 levels | Before product administration and 2, 4, 6 ,8, 10,12, 24 and 48 hours after product administration
  The primary endpoint will be the plasma GDF15 level before and at different timepoints after colchicine administration. Plasma GDF-15 level will be determined using an enzyme immunoassay (EIA) testing.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon request to the principal investigator following the publication of the primary manuscript.